CLINICAL TRIAL: NCT01662011
Title: Application of Neurally Adjusted Ventilatory Assist to Children After Congenital Cardiac Surgery: the Effect of Patient-ventilator Interaction, Gas Exchange and Hemodynamics
Brief Title: Application of Neurally Adjusted Ventilatory Assist to Children After Congenital Cardiac Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Limin Zhu, Attendant doctor, Department of thoracic and cardiovascular surgery, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCMC-2010001
Record Dates: First submitted 2011-08-22; First posted 2012-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Mechanical Ventilation Complication; Congenital Heart Disease
Keywords: patient-ventilator interaction; neurally adjusted ventilatory assist; diaphragm electrical activity; pressure support ventilation
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAVA group (Experimental): Patients ventilated with the mode of neurally adjusted ventilatory assist
  Interventions: Device: mode of neurally adjusted ventilatory assist
- PSV group (Active Comparator): Patients ventilated with the mode of pressure support ventilation.
  Interventions: Device: Mode of pressure support ventilation

INTERVENTIONS:
Device: mode of neurally adjusted ventilatory assist — patients ventilated with the mode of neurally adjusted ventilatory assist after corrective open-heart surgery
  Arms: NAVA group
Device: Mode of pressure support ventilation — Patients ventilated with the mode of pressure support ventilation after corrective open-heart surgery
  Arms: PSV group

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) is a new mode of mechanical ventilation that delivers ventilatory assist in proportion to neural effort. It was a controlled randomized single-center prospective study in order to explore the efficacy of this new mode of mechanical ventilation after corrective open-heart surgery for congenital heart disease.

DETAILED DESCRIPTION:
1. To evaluate the effect of the patient-ventilator interaction in children underwent open-heart surgery when ventilated with NAVA, compared with conventional mechanical ventilation.
2. To verify the benefits of NAVA in improving the gas exchange and hemodynamics after biventricle repair for CHD.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent cardiac surgery with biventricle repaired
* patients need mechanical ventilation more than 24hrs after cardiac surgery

Exclusion Criteria:

* age >18 years
* inappositely of catheter insertion
* hemodynamic instability
* coagulation disorders or bleeding
* inclusion in other research protocol

Ages: 7 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Asynchrony index and Comfort Scale | 2 weeks

SECONDARY OUTCOMES:
Dosage of sedatives | 2 weeks
hemodynamics | 2 weeks
Duration of mechanical ventilation | 2 weeks
Gas exchange | 2 weeks
Length of ICU stay | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Limin Zhu, MD, Study Director — Cardiac intensive care unit, Department of Thoracic and cardiovascular Surgery, Shanghai children's Medical Center
Locations (1):
- Cardiac intensive care unit, Department of cardiothoracic vascular surgery, Shanghai Children's Medical Center, Medical college of Shanghai Jiaotong University, Shanghai, China